CLINICAL TRIAL: NCT02673788
Title: Follow-Up Study of Safety of Pneumostem® in Premature Infants With Intraventricular Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Soon Park, Professor, Samsung Medical Center
Other Study IDs: 2015-09-102
Record Dates: First submitted 2016-01-26; First posted 2016-02-04 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Intracranial Hemorrhages; Mesenchymal Stem Cells; Newborn Infant
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Observation; Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observation without intervention in this follow up study — observation without intervention in this follow up study

SUMMARY:
This is a follow-up study of the open label, single-center, phase I clinical trial to evaluate the safety of Pneumostem® in premature infants with Intraventricular hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Patients who enrolled in the previous phase 1 clinical trial of Pneumostem transplantation for IVH.

Exclusion Criteria:

* Patients who did not enrolled in the previous phase 1 clinical trial of Pneumostem transplantation for IVH.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paitents who enrolled in the previous phase 1 clinical trial of Pneumostem transplantation for IVH.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
newly developed brain tumor | until 2 years old (corrected age)
  Using brain MRI, it is to assess the risk of tumorigenicity of donor stem cells.

SECONDARY OUTCOMES:
Bayley score (MDI, PDI) | until 2 years old (corrected age)
Cerebral palsy | until 2 years old (corrected age)
  more than score 2 based on Gross Motor Function Classification System (GMFCS) score
Developmental disability | until 2 years old (corrected age)
  scoring (category: gait, sitting, hand use, head control, communication, vision, hearing)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No